CLINICAL TRIAL: NCT07290309
Title: Efficacy of a Group-based Videoconference Intervention to Increase Physical Activity in Cancer Survivors
Brief Title: Survivors Uniting for Remote Guided Exercise
Acronym: SURGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Leach, PhD, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6002; 1R01CA296965-01 (NIH)
Record Dates: First submitted 2025-12-15; First posted 2025-12-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cancer (Colon Cancer, Breast Cancer, Lymphoma, Chronic Lymphoma Leukemia, Multiple Myeloma); Physical Activity; Physical Activity Behavior; Cancer (With or Without Metastasis); Cancer - Chronic Lymphocytic Leukemia; Cancer - Ovarian
Keywords: Exercise oncology; Physical activity for cancer survivors; Group based exercise; Virtual exercise; physical activity; exercise; remote study; Cancer survivors
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma; Multiple Myeloma; Motor Activity; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a two-arm randomized controlled trial. Following the NIH Stage Model for Behavioral Intervention Development, we propose a stage II intervention, with the goal of traditional efficacy testing consisting of experimental testing in research settings, with research-based providers
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Virtually Supervised Exercise Class) (Experimental): Live, group-based exercise classes will be delivered 2x per week on Zoom for 12-weeks along with a total of 5 behavior change discussion sessions.
  Interventions: Behavioral: Virtually Supervised Exercise Sessions
- Comparator (Asynchronous Exercise Sessions) (Active Comparator): Participants will watch pre-recorded exercise and discussion videos for 12-weeks.
  Interventions: Behavioral: Asynchronous Group

INTERVENTIONS:
Behavioral: Virtually Supervised Exercise Sessions — The 12-week intervention will consist of supervised exercise sessions twice per week, and PA behavior change discussion sessions twice per month (bi-weekly) throughout the study for a total of five sessions (Week 2, 4, 6, 8 and 10). Exercise and PA behavior change discussion sessions will be informed by social cognitive theory, operationalize several BCT's, and include group dynamics-based strategies to enhance group cohesion. Exercise sessions will take place twice per week, lasting approximately one hour.
  Other Names: Live, Group-Based Zoom Class
  Arms: Intervention (Virtually Supervised Exercise Class)
Behavioral: Asynchronous Group — The comparator will be an "unsupported intervention",128 which will use the same technology and provide the same content as the intervention but subtract the human components. Participants in the control group will receive access to pre-recorded (i.e., asynchronous) videos of the exercise and discussion sessions. The exercise videos will follow the same format as those in the intervention (i.e., instructor led, circuit-style aerobic and resistance exercises). Discussion sessions will operationalize the same BCT's using PowerPoint slides. Comparator arm participants will receive instructions on how to access these videos via a unique participant login to a secure website, Canvas, the same recommendations to achieve PA guidelines, and the same home-based exercise equipment (along with instructions for use).
  Other Names: Pre-recorded exercise videos
  Arms: Comparator (Asynchronous Exercise Sessions)

SUMMARY:
The goal of this research study is to look at how live, online group exercise compares to recorded videos for helping increase physical activity levels, improve physical fitness and quality of life, and reduce loneliness among those living with and beyond cancer. The following aims have been established for this study:

* Aim 1: Examine the effect of a group-based videoconference physical activity (PA) intervention on moderate to vigorous physical activity [MVPA] (i.e., aerobic and resistance exercise).
* Aim 2: Examine the effect of the intervention on additional health-related outcomes including physical fitness (i.e., aerobic endurance, muscular strength), and quality of life at both timepoints.
* Aim 3: Explore potential mediators and moderators of intervention effects. We will examine mediators (e.g., self-efficacy, outcome expectations, group cohesion) and moderators (e.g., age, cancer stage, neighborhood walkability) of the intervention on MVPA.
* Exploratory Aim: Determine whether a group-based videoconference PA intervention reduces loneliness among cancer survivors.

Researchers will randomize participants into one of two guided exercise groups that are 12-weeks long in duration. Participants will be asked to complete online fitness assessments and surveys as well as wear a physical activity monitor device and watch a few times throughout the study. The whole study is 9-months long in duration with a 6-month free-living period where no study activities will take place.

DETAILED DESCRIPTION:
For cancer survivors, moderate to vigorous intensity physical activity (MVPA) is associated with up to 50% reductions in cancer-specific and all-cause mortality. Previous studies also consistently demonstrate that MVPA improves cancer survivor's' physical function and quality of life. However, recent estimates suggest that only 14.2% of cancer survivors engage in the amount of MVPA considered necessary to achieve these health benefits, indicating a need for effective and wide-reaching interventions to increase MVPA.

Supervised interventions that utilize behavior change techniques like goal setting, social support, self-monitoring, action planning, and instruction on how to perform behavior, are most successful in increasing PA among cancer survivors. However, delivering these interventions face-to-face can be resource intensive, and present a barrier to cancer survivors in terms of access (e.g., no programs available nearby, and recently, due to social distancing requirements of the COVID-19 pandemic).

Web, text messaging, and other remote or distance-based PA interventions for cancer survivors demonstrate promise however they exhibit a smaller magnitude of effect on MVPA and physical and psychosocial outcomes than those that are delivered face-to-face. Key factors for this diminished effect size may be lower adherence/compliance due to lack of supervision, and fewer opportunities available for social interaction and support. Cancer survivors acknowledge the importance of peer support for PA, report that one of the quintessential facilitators for engaging in PA is the social benefit and describe camaraderie and the opportunity to be surrounded by others with a shared experience as motivating for being physically active.

The majority of remote or distance-based PA interventions for cancer survivors have been delivered asynchronously (i.e., occurs through online channels without real-time interaction), which eliminates direct supervision from a qualified exercise professional, and presents a challenge for tangible social connections. Conversely, virtually supervised PA interventions (i.e., using videoconferencing) are delivered synchronously, offering the opportunity for real-time supervision and social interaction, while retaining the scalability and reach advantages of remote delivery modalities. However, to date, there have been no large-scale, randomized controlled trials testing the efficacy of a group-based videoconference intervention to increase MVPA in cancer survivors. Videoconferencing can expand the reach of supervised, group-based interventions while potentially enhancing the effects of asynchronous distance-delivered modalities on MVPA, physical, and psychosocial outcomes. Thus, with the substantial, beneficial effects of PA for cancer survivors and the scalability potential of videoconference delivery, findings from this study stand to have high impact not only on the field of PA/exercise for cancer survivorship but can also inform similar interventions and programs for other chronic disease populations.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak/read English,
* Diagnosed with any type of cancer within the last 5 years
* Completed primary or adjuvant treatment (i.e., chemotherapy, radiation therapy, surgery) with no planned treatment within the next nine months. This does not include long-term or chronic therapies such as anti-hormone or targeted therapies (e.g., aromatase inhibitor, androgen deprivation therapy, immunotherapies)

Exclusion Criteria:

* Existing participation in ≥150 minutes per week of at least moderate intensity aerobic exercise
* Known contraindications for non-medically supervised moderate or greater intensity exercise (e.g., uncontrolled hypertension, inability to walk without an assistive device)
* Current or planned participation in another structured program or intervention intended to encourage participation in exercise or physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in accelerometer measured moderate to vigorous physical activity from baseline to 3- and 6-month follow-up | Assessed at baseline, 3-and 6-month follow-up
  MVPA will be compared between the intervention and comparator arm from baseline to post-intervention (primary endpoint) and six-month follow-up.
Change in self-reported moderate-to-vigorous intensity physical activity from baseline to 3 and 6 month follow-up | Assessed at baseline, 3 and 6-month follow-up
  Assessed by Godin Leisure Time Exercise Questionnaire (GLTEQ)

SECONDARY OUTCOMES:
Quality of life will be assessed by a quantitative self-report questionnaire | Assessed at baseline and 3 and 6 month follow-up
  A quality of life survey will be sent at three time points throughout the study: Enrollment, 3-month follow-up, & 6-month follow-up. QOL is assessed on a scale of (1-5) and has different subscales wherein some subscales have a reverse scoring system.
Physical fitness assessed by sit-to-stand and 2-minute step test | Assessed at baseline and 3 and 6 month follow-up
  Participants will complete a total of three study assessments at the following timepoints: Enrollment, 3 -month follow-up, & 6-month follow-up from program completion

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leach, PhD, Principal Investigator — Colorado State University
Locations (1):
- Human Performance Clinical Research Lab, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website where participants can learn more about the study and register interest — https://www.thesurgestudy.org